CLINICAL TRIAL: NCT03226002
Title: Which Nostril Should be Used for Nasotracheal Intubation With Airtraq NT®: the Right or Left? A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Assistant professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: KÜ GOKAEK 2017/71
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Nasotracheal Intubation
Keywords: Airtraq NT; nasotracheal intubation; right; left

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Airtraq NT right nostril (Active Comparator): nasotracheal intubation with Airtraq NT through the right nostril
  Interventions: Device: Airtraq NT
- Airtraq NT left nostril (Active Comparator): nasotracheal intubation with Airtraq NT through the left nostril
  Interventions: Device: Airtraq NT

INTERVENTIONS:
Device: Airtraq NT — channeled video laryngoscope for nasotracheal intubation

SUMMARY:
After Ethics committee approval investigators decided to enroll 40 patients ASA I-II, 18-60 years of age undergoing maxillofascial, oral and double chin surgery to determine which nostril is more suitable for nasotracheal intubation with nasotracheal Airtraq. We primay aimed to compare the glottis visualization time, intubation time and total intubation times.

DETAILED DESCRIPTION:
After Ethics committee approval, investigators decided to enroll 40 pateints ASA I-II, 18-60 years of age undergoing maxillofascial, oral and double chin surgery to determine which nostril is more suitable for nasotracheal intubation with nasotracheal Airtraq. In addition is the 90° anti-clockwise rotation of the tip of the tube helpful to insert the tube into the trachea. Patients were randomized into right and the left nostril groups. After standard anesthesia induction with propofol and fentanyl, rocuronium was used for muscle relaxation. Primary aim of this prospective study was to compare the glottis visualization time, intubation time and total intubation times. The Cormack-Lehane grades, the need for optimization, tube adjustment maneuvers, hemodynamic data, occurrence of epistaxis of the patients were recorded during the process.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* undergoing elective maxillofacial surgery
* dental surgery
* plastic surgery requiring nasotracheal intubation
* ASA I-II

Exclusion Criteria:

* >18 years and > 65 years
* BMI> 35
* ASA III-IV
* fasted patients
* patients do not require nasotracheal intubation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-10 (Actual)

PRIMARY OUTCOMES:
insertion time of the device | 20 seconds
  handling the device till the optimal glottis visualization occurred
nasotracheal intubation time with the device | 30 seconds
  handling the device till the visualization of tracheal tube through the vocal cords
total nasotracheal intubation time with the device | 40 seconds
  handling the device till the confirmation of nasotracheal intubation with end-tidal carbodioxide

SECONDARY OUTCOMES:
optimisation maneuvers during intubation with the device | 20 seconds
  need for optimisation maneuvers during nasotracheal intubation
minor complications related to the device | 40 seconds
  epistaxis, nose pain, bronchospasm

CONTACTS AND LOCATIONS:
Overall Officials: zehra I Arslan, Principal Investigator — Anesthesiology and Reanimation
Locations (1):
- Kocaeli University School of Medicine, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No